CLINICAL TRIAL: NCT00306228
Title: A Randomised Trial to Evaluate the Role of Paclitaxel Eluting Stent and Tirofiban to Improve the Results of Facilitated PCI in the Treatment of Acute ST- Segment Elevation Myocardial Infarction
Brief Title: Role of Tirofiban and the Paclitaxel Eluting Stent in Postfibrinolysis Angioplasty
Acronym: GRACIA3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GRACIA Group (Other)
Collaborators: Spanish Ministry of Health. (Unknown); Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Francisco Fernandez Aviles, Hospital General Universitario Gregorio Maranon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRACIA 3
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Myocardial Infarction
Keywords: ST elevation acute myocardial infarction; Thrombolysis; Early routine percutaneous coronary intervention; tirofiban; paclitaxel
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- bare-metal stent without tirofiban (Active Comparator): implantation of a bare-metal stent with no tirofiban infusion after fibrinolysis
  Interventions: Procedure: Postfibrinolysis percutaneous coronary intervention
- bare-metal stent with tirofiban (Active Comparator): implantation of a bare-metal stent with tirofiban infusion after fibrinolysis
  Interventions: Procedure: Postfibrinolysis percutaneous coronary intervention
- paclitaxel-eluting stent without tirofiban (Active Comparator): implantation of a paclitaxel eluting-stent with no tirofiban after fibrinolysis
  Interventions: Procedure: Postfibrinolysis percutaneous coronary intervention
- paclitaxel-eluting stent with tirofiban (Active Comparator): implantation of a paclitaxel eluting-stent with tirofiban infusion after fibrinolysis
  Interventions: Procedure: Postfibrinolysis percutaneous coronary intervention

INTERVENTIONS:
Procedure: Postfibrinolysis percutaneous coronary intervention — implantation of a bare-metal stent with no infusion of tirofiban 120 minutes after fibrinolysis
  Other Names: Express stents (Boston Scientific, Natick, Massachusetts)
  Arms: bare-metal stent without tirofiban
Procedure: Postfibrinolysis percutaneous coronary intervention — implantation of a bare-metal stent with infusion of tirofiban 120 minutes after fibrinolysis
  Other Names: Express stents (Boston Scientific, Natick, Massachusetts)
  Arms: bare-metal stent with tirofiban
Procedure: Postfibrinolysis percutaneous coronary intervention — implantation of a paclitaxel eluting-stent with no infusion of tirofiban 120 minutes after fibrinolysis
  Other Names: TAXUS stents (Boston Scientific)
  Arms: paclitaxel-eluting stent without tirofiban
Procedure: Postfibrinolysis percutaneous coronary intervention — implantation of a paclitaxel eluting-stent with infusion of tirofiban 120 minutes after fibrinolysis
  Other Names: TAXUS stents (Boston Scientific)
  Arms: paclitaxel-eluting stent with tirofiban

SUMMARY:
The conceptual hypothesis of this study is that, in patients with acute myocardial infarction and ST-segment elevation, the strategy of performing coronary angioplasty of the culprit artery with paclitaxel eluting stent significantly reduces the rate of restenosis in comparison with bare stents.

The conceptual hypothesis of this study is that, in patients with acute myocardial infarction and ST-segment elevation, the strategy of performing coronary stent-angioplasty of the culprit artery under the protection of tirofiban 120 minutes after fibrinolytic significantly improves epicardial and myocardial infusion in comparison with the strategy of performing immediate intravenous thrombolysis (tenecteplase plus enoxaparine) followed by coronary angiography and adequate revascularization.

DETAILED DESCRIPTION:
The primary objectives of this study are: first to determine the efficacy of paclitaxel eluting stent compared to conventional bare stent in terms of restenosis, and second to determine the effect of tirofiban administered prior to percutaneous coronary intervention (PCI) but 120 minutes after thrombolytic on the epicardial and myocardial flow after mechanical revascularization in patients with STEMI.

Methods: This is a phased 4, 2x2 randomised, open, multicenter, clinical study. Patients will be randomised 1:1:1:1 to four groups: a) paclitaxel eluting stent with tirofiban, b) paclitaxel eluting stent without tirofiban, c) bare stent with tirofiban and d) bare stent without tirofiban. A total of approximately 436 patients, with <12 hours STEMI will be enrolled. All patients will be initially treated with tenecteplase (TNK) and enoxaparin. Tirofiban will start 120 minutes after tenecteplase administration in those patients randomised to tirofiban. Cardiac catheterization will be performed within the first 3-12 hours after the study inclusion and stenting on the culprit artery, with the randomised paclitaxel or bare stent, will be performed.

The efficacy of these strategies will be measured in terms of: 1) binary restenosis, defined as >50% diameter stenosis and segment analysis including the stented segment as well as their margins, 5 mm proximal and distal to the stent at 9-12 months follow-up and, 2) the assessment of the epicardial and myocardial perfusion (%TIMI 3, CTFC, CFR-CTFC, TMP y DSA-TMP and the analysis of the normalization of the ST segment at 90 minutes, 3, 6, 12 and 24 hours after thrombolysis).

ELIGIBILITY:
Inclusion Criteria:

Patients with ST-segment elevation acute myocardial infarction with all of the following criteria will be eligible for enrollment:

1. Age >18 years.
2. Chest discomfort >30 minutes with no response to nitroglycerin.
3. Time from the onset of symptoms to randomization < 12 hours.
4. ST segment elevation > 1 mm in two or more limb leads or 2 mm in two or more contiguous precordial leads or non-diagnostic ECG (left bundle branch block or pacemaker rhythm) with classic symptoms.
5. Killip class > 3.
6. Written informed consent will be obtained.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the study.

1. Cardiogenic shock defined as a systolic blood pressure <90 mm Hg without response to fluid administration or <100 mmHg in patients with supportive treatment and no bradycardia.
2. Suspected mechanical complications of acute myocardial infarction.
3. Previous CABG.
4. Non-cardiac disease that is likely to jeopardize the planned termination of the study.
5. Woman of childbearing potential unless a negative pregnant test.
6. Active bleeding and recent (within 2 weeks) surgery that contraindicate the use of heparin, tirofiban, or platelet aggregation inhibitors.
7. Contraindications for thrombolytic use.

   * previous hemorrhagic stroke at any time
   * history of prior non-hemorrhagic cerebrovascular accident within 12 months
   * intracerebral neoplasia
   * active internal bleeding
   * suspected aortic dissection
   * Uncontrolled hypertension >180/110 in several measurements
   * any other known intracerebral pathology not covered in contraindications
   * Current use of anticoagulants or heparin use within 8 hours
   * known bleeding diathesis
   * recent trauma (< 4 weeks), including head trauma or traumatic or prolonged (>10 minutes) CPR or recent major surgery or biopsy (<8 weeks)
   * noncompressible vascular punctures
   * recent (< 4 weeks) internal bleeding
   * pregnancy
   * active peptic ulcer
8. History of hypersensitivity to aspirin, ticlopidine, clopidogrel, heparin, tirofiban and stainless steel.
9. Known renal failure, creatinine >2,5 mg/dL.
10. Known impaired hepatic function that contraindicates the use of clopidogrel.
11. Known thrombocytopenia (100.000).
12. Participation in other trial.
13. Known multivessel disease identified as no suitable for revascularization.
14. Known peripheral vascular disease that difficult cardiac catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2004-10; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
to determine the efficacy of paclitaxel eluting stent compared to conventional bare stent in terms of restenosis | 12 months
to determine the effect of tirofiban administered prior to PCI but 120 minutes after thrombolytic on the epicardial and myocardial flow after mechanical revascularization in patients with STEMI | 24 hours

SECONDARY OUTCOMES:
to determine the safety of paclitaxel eluting stent in terms of rate of complications, and particularly acute and subacute total occlusion. | 12 months
to determine the interaction of paclitaxel eluting stent and the complicated myocardial infarction lesion in terms of reduction of intimal proliferation as evaluated by quantitative coronary angiography | 12 months
to determine the efficacy of paclitaxel eluting stent in different subgroups of patients: diabetics, small vessel (<2.5 mm), long lesion (>15 mm), gender, and tirofiban use. | 12 months
to determine the efficacy and safety of full dose fibrinolytic therapy plus delayed tirofiban compared to fibrinolytic therapy alone in different subgroups: diabetics and the elderly | 30 days
to determine the efficacy of use of tirofiban in relation to time to fibrinolytic therapy and time to mechanical revascularization. | 24 hours
to determine possible interactions between the paclitaxel eluting stent and tirofiban in terms of restenosis or acute and subacute total occlusion following coronary stenting. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fernandez-Aviles, MD, PhD, Study Chair — ICICOR, Hospital Clínico Universitario Valladolid, Spain
Locations (1):
- Instituto de Ciencias del Corazón (ICICOR). Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid, Spain

REFERENCES:
- [Derived] Sanchez PL, Gimeno F, Ancillo P, Sanz JJ, Alonso-Briales JH, Bosa F, Santos I, Sanchis J, Bethencourt A, Lopez-Messa J, de Prado AP, Alonso JJ, San Roman JA, Fernandez-Aviles F. Role of the paclitaxel-eluting stent and tirofiban in patients with ST-elevation myocardial infarction undergoing postfibrinolysis angioplasty: the GRACIA-3 randomized clinical trial. Circ Cardiovasc Interv. 2010 Aug;3(4):297-307. doi: 10.1161/CIRCINTERVENTIONS.109.920868. PMID 20716757